CLINICAL TRIAL: NCT00808717
Title: Efficacy of High Dose Atorvastatin Loading in ST Elevation Myocardial Infarction
Brief Title: Efficacy of High Dose atorvaSTATIN Loading Before Primary Percutaneous Coronary Intervention in ST Elevation Myocardial Infarction (STATIN STEMI)
Acronym: STATIN STEMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Donghoon Choi, Cardiology, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2007-0156
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Myocardial Infarction; Angioplasty; Percutaneous Coronary
Keywords: Myocardial Infarction; Coronary Angioplasty; Myocardial infarction, Angioplasty, Transluminal, Percutaneous Coronary
MeSH Terms: conditions — Myocardial Infarction | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose Atorvastatin 80 mg (Experimental): Administered Atorvastatin 80 mg before intervention
  Interventions: Drug: Atorvastatin
- Control (Active Comparator): Administered Atorvastatin 10 mg before intervention
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 10 mg vs. 80 mg before intervention

SUMMARY:
Although statin prior to PCI has favorable effects in stable angina and ACS except ST elevation MI (STEMI), there have been few studies for STEMI. Celik T et al. reported in patients with STEMI that prior statin use may improve coronary blood flow after PCI in patients with AMI, possibly by its beneficial effects on microvascular function. But this study was retrospective, non-randomized study and evaluated the effects for chronic statin therapy not acute high dose effect. Therefore, the investigators investigated whether acute high-dose statin prior to primary PCI in ST segment elevation myocardial infarction can have beneficial effect or not for periprocedural period and 30 days-cardiac events.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 18 years and 80 years of age.
2. The patient had the symptoms of acute myocardial infarction within 12 hours with ST segment elevation of more than 1 mm in at least two contiguous leads of EKG or new onset LBBB.
3. The patient or guardian agrees to the study protocol and provides informed, written consent.

Exclusion Criteria:

1. Patients to whom PCI can not be undergone within 12 hours from receiving the study drug
2. Cardiogenic shock or symptomatic hypotension or sitting SBP < 95 mmHg
3. The history of major surgery, trauma, retinal hemorrhage, significant gastrointestinal or genitourinary bleeding within recent 6 weeks; history of cerebrovascular attack within two years, or cerebrovascular attack with a significant residual neurological deficit
4. History of cerebrovascular attack within two years, or cerebrovascular attack with a significant residual neurological deficit
5. Severe or malignant hypertension (= sitting SBP > 180 mmHg and/or sitting DBP > 105 mmHg)
6. The history or diagnosis of vasculitis; renal insufficiency (the level of serum creatinine is two times higher than the upper limit of normal of each center)
7. The patients who might die of other disease than cardiac disease during the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of high dose atorvastatin in STEMI - 30 Days MACE(death, myocardial infarction, target vessel revascularization) | 30 days

SECONDARY OUTCOMES:
To evaluate the safety of high dose atorvastatin in STEMI - TIMI flow at before and after PCI - Myocardial blush grade after PCI - Procedural success (No reflow incidence) - MACE at 6 month - Periprocedural MI | immediate, 30 days, 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim JS, Kim J, Choi D, Lee CJ, Lee SH, Ko YG, Hong MK, Kim BK, Oh SJ, Jeon DW, Yang JY, Cho JR, Lee NH, Cho YH, Cho DK, Jang Y. Efficacy of high-dose atorvastatin loading before primary percutaneous coronary intervention in ST-segment elevation myocardial infarction: the STATIN STEMI trial. JACC Cardiovasc Interv. 2010 Mar;3(3):332-9. doi: 10.1016/j.jcin.2009.11.021. PMID 20298994